CLINICAL TRIAL: NCT00764777
Title: Physician Initiated Multi-center Belgian-Italian-Dutch Trial Investigating Abbott Vascular Iliac Stents in the Treatment of TASC A, B, C & D Iliac Lesions
Brief Title: Efficacy Study of Iliac Stents to Treat TASC A-B-C-D Iliac Artery Lesions
Acronym: BRAVISSIMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-006
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Peripheral Vascular Disease; Intermittent Claudication; Critical Limb Ischemia
Keywords: Peripheral Vascular Disease; Intermittent Claudication; Critical limb Ischemia; TASC A; TASC B; TASC C; TASC D; balloon-expandable stent; Self-expanding stent; TASC
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stenting (Experimental)
  Interventions: Device: iliac stenting

INTERVENTIONS:
Device: iliac stenting — Absolute Pro (Abbott Vascular) or Omnilink Elite (Abbott Vascular) stents

SUMMARY:
The BRAVISSIMO trial wants to investigate in a controlled setting, the long-term (up to 24 months) outcome of the self-expanding nitinol Absolute Pro (Abbott Vascular) and the balloon-expandable Omnilink Elite (Abbott Vascular) stent in TASC A&B and TASC C&D iliac lesions. A separate analysis of both patient populations will be performed and listed.

ELIGIBILITY:
Inclusion Criteria:

GENERAL

* Patient presenting with a stenotic or occlusive lesion at the iliac arteries suitable for stenting (on indication for primary stenting, based on the discretion of the investigator)
* Patient presenting a score from 2 to 5 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient is eligible for treatment with the Absolute Pro or Omnilink Elite (Abbott Vascular)

ANGIOGRAPHIC

* The target lesion is either a modified TASC-II class A, B, C or D lesion with one of the listed specifications:
* Type A lesions
* Unilateral or bilateral stenoses of the Common Iliac Artery
* Unilateral or bilateral single short (≤3 cm) stenosis of the External Iliac Artery
* Type B lesions
* Unilateral Common Iliac Artery occlusion
* Single or multiple stenosis totaling 3-10 cm involving the External Iliac Artery not extending into the Common Femoral Artery
* Unilateral External Iliac Artery occlusion not involving the origins of Internal Iliac Artery or Common Iliac Artery
* Type C lesions
* Bilateral Common Iliac Artery occlusions
* Bilateral External Iliac Artery stenoses 3-10 cm long not extending into the Common Femoral Artery
* Unilateral External Iliac Artery stenosis extending into the Common Femoral Artery
* Unilateral External Iliac Artery occlusion that involves the origins of the Internal Iliac and/or Common Femoral Artery
* Heavily calcified unilateral External Iliac Artery occlusion with or without involvement of origins of the Internal Iliac and/or Common Femoral Artery
* Type D lesions
* Unilateral occlusions of both Common Iliac and External Iliac Artery
* Diffuse disease involving the aorta and both iliac arteries requiring treatment
* Diffuse multiple stenoses involving the unilateral Common Iliac, External Iliac and Common Femoral Artery
* Bilateral occlusions of External Iliac Artery
* The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
* There is angiographic evidence of a patent Common an Deep Femoral Artery

Exclusion Criteria:

* The target lesion is either a modified TASC-II class B or D lesion with aortic lesion involvement:
* Type B lesions
* Short (≤3 cm) stenosis of infrarenal aorta
* Type D lesions
* Infra-renal aortoiliac occlusion
* Iliac stenoses in patients with an Abdominal Aortic Aneurysm (AAA) requiring treatment and not amenable to endograft placement or other lesions requiring open aortic or iliac surgery
* Presence of aneurysm at the level of the iliac arteries
* Previously implanted stent(s) at the same lesion site
* Reference segment diameter is not suitable for available stent design
* Untreatable lesion located at the distal outflow arteries
* Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index procedure
* Patients refusing treatment
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with a history of prior life-threatening contrast medium reaction
* Patients with known hypersensitivity to nickel-titanium
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary patency defined as a target lesion without a hemodynamically significant stenosis on duplex ultrasound (>50%, systolic velocity ratio no greater than 2.0) and without TLR | 12 months

SECONDARY OUTCOMES:
Technical success, defined as the ability to achieve final residual angiographic stenosis no greater than 30% | Procedure
Primary patency rate at different follow-up times defined as absence of hemodynamically significant stenosis at the target area on duplex ultrasound (>50%, systolic velocity ratio no greater than 2.0) and without prior TLR. | 1, 6 & 24 months
3) Clinical success at follow-up is defined as an improvement of Rutherford classification at different follow-ups of one class or more as compared to the pre-procedure Rutherford classification. | 1, 6, 12 & 24 months
Serious adverse events | 1, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — AZ Sint-Blasius, Dendermonde, Belgium
Locations (5):
- Belgium (5):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - ZOL Campus Sint-Jan, Genk
  - University Hospital, Ghent